CLINICAL TRIAL: NCT00100581
Title: An Open-Label, Randomized Study to Determine the Impact of Antiretroviral Treatment in HCV/HIV-Coinfected Subjects With High CD4+ Cell Count on the Efficacy of Hepatitis C Treatment With Pegylated Interferon Alfa-2A and Ribavirin
Brief Title: Effects of Anti-HIV Therapy on Treatment for Hepatitis C in HCV/HIV Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5184; 10133 (Registry Identifier: DAIDS ES Registry Number); ACTG A5184
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — efavirenz; Lamivudine; Lopinavir; peginterferon alfa-2a; Ribavirin; Tenofovir

INTERVENTIONS:
Drug: Efavirenz
Drug: Lamivudine
Drug: Lopinavir/ritonavir
Drug: Pegylated interferon alfa-2a
Drug: Ribavirin
Drug: Tenofovir disoproxil fumarate

SUMMARY:
A significant proportion of HIV infected people in the U.S. are also infected with hepatitis C virus (HCV). The purpose of this study is to determine the effects of anti-HIV therapy on treatment of HCV with pegylated interferon alfa-2a and ribavirin (PEG/RBV).

DETAILED DESCRIPTION:
An estimated 15% to 30% of HIV infected people in the U.S. are also infected with HCV. Since the introduction of antiretroviral therapy (ART) for the treatment of HIV, HCV infection has emerged as a major cause of morbidity and mortality in HCV/HIV coinfected patients. One infection often accelerates the progression of the other, and effective management strategies for both infections need to be developed for HCV/HIV coinfected patients. This study will determine whether HIV ART followed by HCV therapy taken concurrently with ART results in better treatment outcomes compared to HCV therapy alone.

This study will last up to 102 weeks. Participants will be randomly assigned to one of two arms. Arm A participants will receive 24 to 30 weeks of ART consisting of tenofovir disoproxil fumarate (TDF) and lamivudine (3TC) and either efavirenz (EFV) or lopinavir/ritonavir (LPV/r). If deemed eligible, Arm A participants will continue their ART regimen and begin a concurrent PEG/RBV regimen for up to 48 weeks. At Week 48, participants in Arm A will stop PEG/RBV and will be followed for an additional 24 weeks on ART alone.

Arm B participants will receive PEG/RBV alone for up to 48 weeks. At Week 48, participants in Arm B will be followed for an additional 48 weeks with no treatment.

There will be 20 study visits over 102 weeks for Arm A participants and 18 study visits over 96 weeks for Arm B participants. Blood collection and clinical assessment will occur at all visits, and urine collection will occur at selected visits. Participants will also be asked to complete adherence questionnaires. Participants in this study are encouraged to also enroll in ACTG A5128.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV infected
* HIV viral load of greater than 1000 copies/ml within 45 days of study entry
* HCV genotype 1 infected
* CD4 count of 300 cells/mm3 or greater within 45 days prior to study entry
* ART-naive or off ART for at least 6 months
* Willing to accept randomly assigned study treatment
* Willing to use acceptable forms of contraception during the study and for 6 months after stopping all study medications
* Chronic liver disease consistent with chronic viral hepatitis as indicated by either liver biopsy within 2 years prior to study entry or a physician's report of hepatitis C infection for more than 6 months. Participants with cirrhosis or without a liver biopsy result within 2 years of study entry must have a serum alpha-fetoprotein of 100 ng/ml or less and a Child-Pugh score of 6 or higher within 45 days prior to study entry to be eligible for this study.

Exclusion Criteria for Step 1:

* Hepatitis B surface antigen positive within 45 days prior to study entry
* HCV genotype other than genotype 1 at any time prior to study entry
* Any medical conditions associated with chronic liver disease other than HCV (e.g., genetic hemochromatosis, autoimmune hepatitis)
* Prior use of intravenous or subcutaneous interferon for more than 2 weeks total at any time prior to study entry
* Known allergy/sensitivity to pegylated interferon alpha-2a, ribavirin, or their formulations
* Current drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study. Participants in methadone programs are not excluded, but may require methadone dose changes during the study.
* Need to start ART at the time of study entry
* Uncontrolled diabetes mellitus within 30 days prior to study entry
* Previous suicide attempt or hospitalization for a psychiatric illness within 6 months prior to study entry. Participants with psychiatric disease, especially depression, uncontrolled with medication are not eligible for the study.
* Prior or current evidence of immunologically mediated disease (e.g., inflammatory bowel disease, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis)
* Chronic pulmonary disease associated with functional limitation
* Severe cardiac disease within 24 weeks prior to study entry
* History of severe retinopathy due to diabetes, hypertension, cytomegalovirus, or macular degeneration
* History of major organ transplantation
* Severe illness, cancer, or other conditions that would interfere with the study
* Any systemic antineoplastic or immunomodulatory treatment (except epoetin alfa or granulocyte colony-stimulating factor [G-CSF]) or radiation within 24 weeks of study entry. Participants who anticipate the need to begin such treatment during the study are not eligible.
* History of hemoglobinopathy (e.g., thalassemia, sickle cell anemia)
* Require certain medications
* Evidence of decompensated liver disease, such as history or presence of ascites, jaundice, bleeding varices, or hepatic encephalopathy
* Prior opportunistic infection or lowest ever CD4 count less than 200 cells/mm3
* Has a pregnant partner
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
HCV viral load at least 2 log10 less than baseline or below the limit of detection by quantitative assay at 12 weeks after the start of HCV treatment (early virologic response)
HIV and/or HCV treatment-limiting or Grade 4 or higher signs and symptoms and laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gripshover, MD, Study Chair — University Hospitals of Cleveland, Case Western Reserve University; Mark S. Sulkowski, MD, Study Chair — Viral Hepatitis Center, Johns Hopkins University School of Medicine
Locations (2):
- United States (2):
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas

REFERENCES:
- [Background] Mehta SH, Thomas DL, Torbenson M, Brinkley S, Mirel L, Chaisson RE, Moore RD, Sulkowski MS. The effect of antiretroviral therapy on liver disease among adults with HIV and hepatitis C coinfection. Hepatology. 2005 Jan;41(1):123-31. doi: 10.1002/hep.20541. PMID 15619237
- [Background] Plosker GL, Keating GM. Peginterferon-alpha-2a (40kD) plus ribavirin: a review of its use in hepatitis C Virus And HIV co-infection. Drugs. 2004;64(24):2823-43. doi: 10.2165/00003495-200464240-00009. PMID 15563253
- [Background] Sterling RK, Sulkowski MS. Hepatitis C virus in the setting of HIV or hepatitis B virus coinfection. Semin Liver Dis. 2004;24 Suppl 2:61-8. doi: 10.1055/s-2004-832930. PMID 15346248
- [Background] Sulkowski MS, Moore RD, Mehta SH, Chaisson RE, Thomas DL. Hepatitis C and progression of HIV disease. JAMA. 2002 Jul 10;288(2):199-206. doi: 10.1001/jama.288.2.199. PMID 12095384
- [Background] Sulkowski MS, Thomas DL. Hepatitis C in the HIV-infected patient. Clin Liver Dis. 2003 Feb;7(1):179-94. doi: 10.1016/s1089-3261(02)00074-0. PMID 12691466
- See also: Click here for more information on ACTG A5128 — http://clinicaltrials.gov/ct/show/NCT00031408